CLINICAL TRIAL: NCT06389734
Title: The Effects of Combining Manual Soft Tissue Release and Physical Exercise Training on Lung Function(LF), Exercise Capacity(EC), and Cardiac Autonomic Function(CAF) in Moderate to Severe COPD: A Randomized Controlled Trial
Brief Title: Combining Manual Soft Tissue Release and Exercise Training in COPD: the Effect on LF, EC, and CAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Kun-Ling Tsai, Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B-ER-111-470
Record Dates: First submitted 2024-04-15; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Manual Soft Tissue Release; Exercise Training; Lung Function; Exercise Capacity; Cardiac Autonomic Function
Keywords: chronic obstructive pulmonary disease; manual soft tissue release; exercise training; lung function; exercise capacity; cardiac autonomic function; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Myofascial Release Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: The study population will be randomized and separated in two groups, experimental and control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive combining manual soft tissue release and exercise training.
  Interventions: Behavioral: Manual soft tissue release; Behavioral: Exercise training
- Control group (Active Comparator): The control group will receive combining myofascial release and exercise training.
  Interventions: Behavioral: Myofascial release; Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Manual soft tissue release — The manual soft tissue release includes muscle energy techniques and passive stretching, targeting the anterior scalene, upper trapezius, pectoralis major, pectoralis minor, and diaphragm.
  Three times a week for six weeks, with three rounds per session, each session having three repetitions, with a 30-second break in between, lasting 15 to 30 seconds each time.
  Arms: Intervention group
Behavioral: Myofascial release — The myofascial release includes suboccipital muscle, anterior chest wall myofascial, and anterior neck myofascial.
  Three times a week for six weeks, with three rounds per session, each session having three repetitions, with a 30-second break in between, lasting 15 to 30 seconds each time.
  Arms: Control group
Behavioral: Exercise training — The exercise training includes aerobic exercise training by treadmill. The initial intensity is set at 60% to 85% of the average speed measured during the patient's six-minute walk test (6MWT). Intensity adjustments will be made using the Modified Borg Scale (scores ranging from 4 to 7). Training duration is 30 minutes, three times a week for six weeks.

SUMMARY:
The potential effects of combining manual soft tissue release and physical exercise training on lung function, exercise capacity, and cardiac autonomic function in patients with moderate and severe chronic obstructive pulmonary disease were investigated.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) commonly presents with accessory respiratory muscle tightness and weakness, affecting chest wall compliance and lung elasticity. However, traditional physical therapy interventions, including pursed-lip breathing, sputum clearance techniques, and respiratory muscle training, are often used in treatment guidelines, with few studies focusing on muscle release for the accessory respiratory muscles. Although the effects of manual therapy on lung function and chest tightness in COPD have been demonstrated, the effects of soft tissue release combined with exercise intervention on COPD, including lung function, exercise capacity, and cardiac autonomic function, remain unknown. Therefore, this study proposes a randomized controlled trial to investigate the effects of manual soft tissue release combined with exercise training on lung function, exercise capacity, and cardiac autonomic function in patients with COPD. It is expected that the results of this study will demonstrate that combining manual soft tissue release with exercise training may increase gas exchange in the lungs, reduce respiratory effort, improve co-morbidities, delay disease progression, and enhance patient quality of life and clinical intervention.

ELIGIBILITY:
Inclusion Criteria:

* GOLD grade II~IV
* Stable condition
* No acute exacerbations in 6 weeks

Exclusion Criteria:

* Acute heart failure and, or arrhythmia
* Pulmonary arterial hypertension
* Skeletal and, or neuromuscular disorders
* Chest surgery
* Untreated or uncontrolled conditions
* Rheumatoid conditions
* Depends on oxygen supply

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 s (FEV1) | Change from baseline (0 week) to follow-up (12 weeks)
  FEV1 is measured by the lung function test, and the unit presented will be in percent and liter.
forced vital capacity (FVC) | Change from baseline (0 week) to follow-up (12 weeks)
  FVC is measured by the lung function test, and the unit presented will be in percent and liter.
FEV1/FVC ratio | Change from baseline (0 week) to follow-up (12 weeks)
  FEV1/FVC ratio is measured by the lung function test, and the unit presented will be in percent.
expiratory reserve volume (ERV) | Change from baseline (0 week) to follow-up (12 weeks)
  ERV is measured by the lung function test, and the unit presented will be in liter.
functional residual capacity (FRC) | Change from baseline (0 week) to follow-up (12 weeks)
  FRC is measured by the lung functions test, and the unit presented will be in liters.
inspiratory capacity (IC) | Change from baseline (0 week) to follow-up (12 weeks)
  IC is measured by the lung functions test, and the unit presented will be in liters.
inspiratory reserve volume (IRV), | Change from baseline (0 week) to follow-up (12 weeks)
  IRV is measured by the lung functions test, and the unit presented will be in liters.
residual volume (RV) | Change from baseline (0 week) to follow-up (12 weeks)
  RV is measured by the lung function test, and the unit presented will be in liters.
total lung capacity (TLC) | Change from baseline (0 week) to follow-up (12 weeks)
  TLC is measured by the lung function test, and the unit presented will be in liters.
tidal volume (TV) | Change from baseline (0 week) to follow-up (12 weeks)
  TV is measured by the lung function test, and the unit presented will be in liters.
vital capacity (VC) | Change from baseline (0 week) to follow-up (12 weeks)
  VC is measured by the lung function test, and the unit presented will be in liters.

SECONDARY OUTCOMES:
Rate of perceived exertion (RPE) | Change from baseline (0 week) to follow-up (12 weeks)
  RPE is measured by the cardiopulmonary exercise test. This scale ranges from 0 (very light activity) to 10 (maximum effort activity).
Oxygen consumption (VO2) | Change from baseline (0 week) to follow-up (12 weeks)
  VO2 is measured by the cardiopulmonary exercise test, and the unit presented will be in milliliters of oxygen consumed per minute (ml/min).
oxygen saturation | Change from baseline (0 week) to follow-up (12 weeks)
  oxygen saturation is measured by the oximeter, and the unit presented will be in percent
heart rate (HR) | Change from baseline (0 week) to follow-up (12 weeks)
  HR is measured by cardiopulmonary exercise test, and the unit presented will be in beat per minute (BPM)
blood pressure (BP) | Change from baseline (0 week) to follow-up (12 weeks)
  BP is measured by the cardiopulmonary exercise test, which is divided into two parameters: systolic blood pressure (SBP) and diastolic blood pressure (DBP).
  The unit presented will be in millimeters of mercury (mmHg).
Diaphragmatic mobility | Change from baseline (0 week) to follow-up (12 weeks)
  Diaphragmatic mobility is measured by the ultrasound, and the unit presented will be in millimeters
Cardiac Autonomic Function | Change from baseline (0 week) to follow-up (12 weeks)
  Cardiac Autonomic Function is measured by heart rate variability of electrocardiography, and the unit presented will be in millisecond (ms) and millisecond square (ms2)
six minute walk test (6-MWT) | Change from baseline (0 week) to follow-up (12 weeks)
  6-MWT assesses the distance a person can walk within 6 minutes, and the unit presented will be in meters.
maximal expiratory pressure (MEP) | Change from baseline (0 week) to follow-up (12 weeks)
  MEP is measured by the pressure meter, and the unit presented will be in centimetre of water (cmH2O).
maximal inspiratory pressure (MIP) | Change from baseline (0 week) to follow-up (12 weeks)
  MIP is measured by the pressure meter, and the unit presented will be in centimetre of water (cmH2O).
St. George's Respiratory Questionnaire (SGRQ) | Change from baseline (0 week) to follow-up (12 weeks)
  SGRQ is assessing how obstructive airway disease affects overall health, daily life, and well-being. Scores range from 0 to 100, with higher scores indicating more limitations.
fatigue severity scale (FSS) | Change from baseline (0 week) to follow-up (12 weeks)
  FSS is assessing the impact of fatigue on a person's activity and lifestyle. There are nine items, and each item is scored from 1 to 9 (strongly disagree to strongly agree).
  Higher total scores indicate more severe fatigue.
Modified Medical Research Council (mMRC) | Change from baseline (0 week) to follow-up (12 weeks)
  mMRC is assessing the subjective degree of breathlessness by patients during physical activity. It rates on a scale from 0 to 4, with a higher rate indicating the worst possible shortness of breath.
36-Item Short Form Health Survey (SF-36) | Change from baseline (0 week) to follow-up (12 weeks)
  SF-36 is assessing the subjective survey health status and quality of life. It consists of eight sections, with scores ranging from 0 to 100. Higher scores indicate better health and less disability.

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ling Tsai, Ph.D., Principal Investigator — Study Principal Investigator
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No